CLINICAL TRIAL: NCT03075826
Title: A Phase II Study of SGI-110 in Philadelphia-Negative Myeloproliferative Neoplasms
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Astex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1510016613
Record Dates: First submitted 2017-03-03; First posted 2017-03-09 (Actual); Results first posted 2022-04-06 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-04

CONDITIONS: Myeloproliferative Neoplasms
MeSH Terms: conditions — Myeloproliferative Disorders | interventions — guadecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open Label-Single Arm (Other): This is a single arm, open-label study of SGI-110 in patients with MPN. SGI-110 will be administered subcutaneously at a dose of 60 mg/m2 on days 1-5, repeated every 28 days. Toxicity will be evaluated using the NCI Common Terminology Criteria for Adverse Events Active Version 4. The frequency of toxicities per organ system will be tabulated using descriptive statistics. All patients who receive any amount of the study drug will be evaluable for toxicity
  Interventions: Drug: SGI-110

INTERVENTIONS:
Drug: SGI-110 — subcutaneously at a dose of 60 mg/m2
  Other Names: Guadecitabine

SUMMARY:
* This is an open label single-arm, single-institution stud to evaluate the efficacy and safety of SGI-110 in Philadelphia chromosome negative (Ph-) Myeloproliferative Neoplasms (MPN) (excluding PV, ET and primary/secondary myelofibrosis). The study will enroll approximately 50 patients at the Weill Cornell Medical College.
* Enrollment onto this clinical study is expected to be completed in approximately 36 months. The total study duration will depend on individual response, evidence of disease progression and tolerance. Participants will be followed monthly for six months after removal from study or until death, whichever occurs first.

Key eligibility:

* Confirmed diagnosis of Ph- MPN and had
* No chemotherapy or radiation treatment within 2 weeks prior to study entry.
* Subjects meet other protocol-defined criteria related to baseline screening procedures.

DETAILED DESCRIPTION:
The active metabolite of SGI-110 (2'-deoxy-5-azacytidylyl-(3'→5')-2'-deoxyguanosine sodium salt), a dinucleotide, is decitabine, an FDA-approved agent for the treatment of myelodysplastic syndromes. SGI-110 is resistant to modification by cytidine deaminase, a common pathway of decitabine metabolism and deactivation[1]. The molecular weight of SGI-110 and decitabine are 580 Da and 228 Da, respectively. Therefore, the molar equivalent dose of 1 mg of decitabine is approximately 2.5 mg of SGI-110. SGI-110's activity was demonstrated with the same preclinical pharmacodynamic assays used to demonstrate decitabine's efficacy e.g., re-expression of p15, p16, and MLH1 and induction of fetal hemoglobin, in vivo. In xenograft studies, SGI-110 demonstrates promising preclinical activity in both hematologic and solid tumors.

In vitro evidence suggests that SGI-110 has a longer half-life than decitabine in the presence of cytidine deaminase. These promising observations suggest that SGI-110 may have improved pharmaceutical properties and biological activities that could extend decitabine's current clinical utility. SGI-110 has shown to be better tolerated in mice than decitabine and is as effective in vivo in inducing p16 expression, reducing DNA methylation at the p16 promoter region, and retarding EJ6 human bladder cancer tumor growth in athymic mice[2].

SGI-110 has been developed for subcutaneous administration. SGI-110 is pharmacologically active both in vitro and in vivo in a variety of tumor cells and murine xenograft models when administered subcutaneously. Treatment is well tolerated via the subcutaneous route in murine xenografts. When administered subcutaneously to non-human primates, SGI-110 releases decitabine slowly compared to other species, possibly prolonging the effect over longer periods. SGI-110 has been developed as a non-aqueous formulation to ensure formulation stability.

SGI-110 has been studied in a first-in-human, single-agent study (SGI-110-01).5 This study was a Phase 1/2, dose escalation, multicenter study of two subcutaneous regimens of SGI-110 in subjects with intermediate or high-risk myelodysplastic syndromes (MDS) or acute myeloid leukemia (AML). This study had two parts, a Dose Escalation Segment and a Dose Expansion Segment. The study evaluated the biological activity, preliminary safety, and efficacy of SGI-110 with two dosing schedules in intermediate to high risk MDS or relapsed or refractory AML subjects, while the Dose Expansion Segment further evaluated safety and efficacy at the recommended dose. The study was based on a 3 + 3 design within each regimen. Eligible subjects were randomized to receive 1 of 2 dosing regimens of SGI-110 with the following starting doses: Regimen 1: 3 mg/m2/day subcutaneously on Days 1-5 of a 28-day course, Regimen 2: 6 mg/m2 subcutaneously Weekly x 3 on Days 1, 8, 15 of a 28-day course. The minimum dose achieving maximal biological activity or biologically effective dose (BED) for the daily regimen was reached at 60 mg/m2 daily on Days 1-5.

Study disease: MPN

Philadelphia chromosome negative Myeloproliferative Neoplasms (PHN-MPN) comprise a group of myeloid neoplasms with varying clinical, morphologic and laboratory features and a wide range of survival. According to 2008 World Health Organization (WHO) classification, the MDS/MPN overlap syndromes include chronic myelomonocytic leukemia (CMML), atypical chronic myeloid leukemia (aCML), juvenile myelomonocytic leukemia(JMML) and myelodysplastic/myeloproliferative neoplasm unclassifiable (MDS/MPN-U). In a recent retrospective study from MD Anderson Cancer Center, the median survival of patients with a diagnosis of MDS/MPN unclassifiable was 12.4 months[3] .There is no effective therapy for PHN-MPN and this represents an unmet medical need.

The MDS/MPN overlap syndromes can present with a wide range of hematological and clinical manifestations and individual patients may exhibit a combination of features characteristic of both MDS and MPN. For example, while transfusion-dependent anemia is generally present, other hematological laboratory abnormalities can range from leukopenia to leukocytosis and from thrombocytopenia to thrombocytosis. Unlike with MDS, significant splenomegaly is often present in patients with PHN-MPN. Also, patients may have a constellation of constitutional findings, including fatigue, weight loss, anorexia, night sweats and other unpleasant symptoms that lead generally to poor quality of life. Thus, while improving overall survival is a critical goal of therapy, effective therapy for this group of patients will include also agents that can be demonstrated to improve as many of the disease-related clinical issues as possible.

Overall Study Design

This is a single arm, open-label study of SGI-110 in patients with MPN. SGI-110 will be administered subcutaneously at a dose of 60 mg/m2 on days 1-5, repeated every 28 days. Toxicity will be evaluated using the NCI Common Terminology Criteria for Adverse Events Active Version 4. The frequency of toxicities per organ system will be tabulated using descriptive statistics. All patients who receive any amount of the study drug will be evaluable for toxicity.

Screening and pre-treatment criteria Screening Procedures Screening procedures and tests will be performed within 14 days before treatment administration with the exception of informed consent, bone marrow biopsy which may be performed within 28 days of the first dose of study drug.

* Provision of written informed consent. The ICF must be signed and dated by the subjects before collection of any samples or performance of any study-specific evaluations.
* Complete medical history, including demographics (date of birth, sex, race). A disease history, including the date of initial diagnosis and list of prior treatments and responses to these treatments, also will be recorded. Concurrent medical signs and symptoms must be documented to establish baseline conditions.
* Record concomitant medications.
* Record all study-procedure related AEs from the time of informed consent and then treatment-emergent AEs after the start of study drug administration (Course 1, Day 1) through 30 days after the last dose of study drug.
* Investigator's confirmation of eligibility. Perform all necessary procedures and evaluations to document that the subject meets each eligibility criterion.
* Complete physical exam including weight and examination
* Vital signs include resting systolic/diastolic blood pressure, resting heart rate, resting respiration rate, body temperature and pulse oximetry. Assess after the subject has rested in the sitting position for at least three minutes.
* ECOG performance status.
* 12-lead ECG (rhythm, atrial rate, ventricular rate, PR interval, QRS duration, and QT/QTc (QtcF), morphology and overall interpretation).
* Height.
* Sample collection for clinical laboratory tests (hematology, chemistry and urinalysis).
* Serum or urine pregnancy test: for female subjects of child-bearing potential only. Results must be negative for the subject to be eligible for enrollment into the study.

Agent Administration

• SGI-110 administered at dose level of 60 mg/m2 SC daily on Days 1-5 of a 28-day cycle. However, treatment delays are allowed per section 6.3.1 SGI-110 is administered by SC injection preferably in the abdominal area. The total amount (in mg) of SGI-110 to be administered will be determined based on the body surface area (BSA). In calculating the BSA, actual heights and weights should be used. There will be no adjustments to "ideal" body weight. The institutional standard for calculating BSA is acceptable. Dose adjustment should be made for a +/- 10% weight change at the beginning of each cycle The site(s) of SGI-110 SC injections will be captured on the dosing CRF. Investigators are prohibited from supplying SGI-110 to any subjects not properly enrolled in this study or to any physicians or scientists except those designated as sub-investigators on Food and Drug Administration (FDA) Form 1572. The investigator must ensure that subjects receive SGI-110 only from personnel who fully understand the procedures for administering the study treatment.

Duration of Therapy

Duration of therapy will depend on individual response, evidence of disease progression and tolerance. In the absence of treatment delays due to adverse events, treatment may continue until one of the following criteria applies:

* Disease progression to acute leukemia unless, in the opinion of the principal investigator, the subject is experiencing clinical benefit from SGI-110 despite laboratory evidence of progression to acute leukemia.
* Intercurrent illness that prevents further administration of treatment,
* Unacceptable adverse event(s)
* Participant demonstrates an inability or unwillingness to comply with the medication regimen and/or documentation requirements
* Participant decides to withdraw from the study
* General or specific changes in the participant's condition render the participant unacceptable for further treatment in the opinion of the treating investigator.

Duration of Follow Up

Participants will be followed monthly for six months after removal from study or until death, whichever occurs first. Participants removed from study for unacceptable adverse events will be followed until resolution or stabilization of the adverse event. Post-study case report forms will capture information including subsequent treatments, response to subsequent therapy, and survival.

Anticipated Toxicities

Adverse Event List(s) for SGI-110

The most common AEs suspected by the investigators in Study SGI-110-01 to be related to the drug and observed to date in the MDS/AML population are: injection site pain, fatigue, nausea, thrombocytopenia, anemia and diarrhea. Based on the mechanism of action of the drug and its active form decitabine, myelosuppression (neutropenia, thrombocytopenia, and anemia) and the related consequences such as infection (e.g. pneumonia), sepsis, and bleeding are the most likely risks for the drug. Mucositis has also been reported.

Pain and burning at the injection site has been reported that are related to dose and volume of injection as well as the speed of injection. Care must be taken to avoid intradermal injection. Ice packs will be applied prior to injection of SGI-110 and the drug will be injected slowly, over 30-60 seconds. If the injection site events are reported at subsequent injections despite slow injection and the use of ice packs, pre-treatment with topical or systemic analgesics can be considered.

ELIGIBILITY:
Inclusion Criteria:

3.1.1 Participants must have confirmed diagnosis of Philadelphia chromosome negative MPN neoplasm based on WHO classification (reference) including Chronic Neutrophilic Leukemia (CNL), atypical Chronic Myeloid Leukemia (aCML), Chronic Myelomonocytic Leukemia (CMML), MPN/MDS overlap syndromes, accelerated phase myelofibrosis and MPN unclassifiable.

3.1.2 Age minimum of 18 years. Because no dosing or adverse event data are currently available on the use of SGI-110 in participants <18 years of age, children are excluded from this study but may be eligible for future pediatric trials.

3.1.3 ECOG performance status <3

3.1.4 Participants must have normal organ function as defined below:

* Total bilirubin < or = 1.5 X institutional upper limit of normal unless attributable to underlying disease, hemolysis or documented Gilbert's syndrome
* AST (SGOT)/ALT (SGPT) < 2.5 X institutional upper limit of normal unless attributable to underlying disease
* Creatinine < 1.5add < or = 1.5X institutional upper limit of normal or creatinine clearance add using Cockcroft Gault > 50 mL/min/1.73 m2 for subjects with creatinine levels above institutional normal.
* LVEF < 40 % is allowed as long as there is no NY class III/IV heart failure or uncontrolled arrhythmias.

3.1.5 The effects of SGI-110 on the developing human fetus are unknown. For this reason and because oncological agents are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

3.1.6 Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

3.2.1 Participants who have had any chemotherapy (investigational or FDA approved) (hydroxyurea is permitted) or radiotherapy within 2 weeks prior to study entry or those who have not recovered from adverse events due to agents administered more than 2 weeks earlier.

3.2.2 Participants may not be treated with any other investigational agents while on this study unless approved by the principal investigator AND the sponsors of BOTH investigational agents.

3.2.3 History of allergic reactions attributed to compounds of similar chemical or biologic composition to decitabine or SGI-110.

3.2.4 Uncontrolled intercurrent illness including, but not limited to, infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Pregnant women are excluded from this study because SGI-110 is a hypomethylating agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk of adverse events in nursing infants secondary to treatment of the mother with SGI-110, breastfeeding should be discontinued.

3.2.5 Individuals with a history of a different malignancy are ineligible except for the following circumstances. Individuals with a history of other malignancies are eligible if they have been disease-free for at least 3 years and are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers are eligible if diagnosed and treated within the past 3 years: cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-03-15 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pinkal Desai, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 22 subjects were treated with SGI-110. Of the 22 that were treated 16 were evaluable for response to study drug.
Period: Overall Study
Arm/Group | Open Label-Single Arm
Started | 22
Completed | 16
Not Completed | 6
Not completed — Withdrawal by Subject | 1
Not completed — Received less than 3 cycles of study drug | 5

BASELINE CHARACTERISTICS:
Arm/Group | Open Label-Single Arm
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Hematological Response, as Measured by Any One or More of the Following Response Assessments: IWG-MDS and IWG-MF Criteria as Accurate and Appropriate.
Description: The response to treatment will be measured from baseline through 12 cycles. A response assessment will be performed after cycle 3, cycle 6 and cycle 12. The response will be measured by IWG-MDS (International working group - Myelodysplastic Syndrome), which is a set of criteria that dictates what response a patient with MDS has had to a treatment; IWG-MF (International Working Group - Myelofibrosis) which is a set of criteria that dictates what response a patient with MF has had to a treatment. Both sets of criteria utilize the following parameters to asses response: Results from blood tests; bone marrow biopsies; physical exams to look at spleen and liver size; and symptoms. All responses will be recorded in our database and the best response to treatment will be reported. A cycle is at least 28 days, which can be extended past day 28 in order to allow physicians decision to delay next cycle based on the patients clinical needs.
Time Frame: At the end of cycles 3, 6 and 12 - up to approximately 336 days
Population: 6 patients were inevaluable - 1 patient withdrew consent and 5 patients received less than 3 cycles of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label-Single Arm
Number analyzed (Participants) | 16
Participants
  Complete remission | 2
  Partial remission | 0
  Complete cytogenetic remission | 0
  Marrow response | 3
  Clinical benefit | 2
  Stable disease | 9

2. Secondary Outcome: Number of Participants With Change in Quality of Life (QoL) Scores as Defined by Myeloproliferative Neoplasms Symptoms Assessment Form (MPN-SAF).
Description: Symptom improvement response is defined as a number of subjects with improvement in symptoms response as defined by Myeloproliferative Neoplasms Symptoms Assessment Form (MPN-SAF). The MPN-SAF is a questionnaire that measures certain symptoms and how they improve throughout the study, from baseline. The questionnaire is divided into 4 sections - 1: 16 questions about the most common symptoms in these disease types, rated from 0 (lowest impact) to 10 (biggest impact); 2: Highest grade of fever; 3: Unintentional weight loss; 4. Quality of life, rated from 0 (as good as it can be) to 10 (as bad as it can be).
Time Frame: Baseline, at the beginning of each new cycle - approximately every 28 days for up to 700 days
Population: Out of 22 patients treated, 21 patients were analyzed for at least one section of the MPN-SAF questionnaire (1 patient came off treatment after 1 cycle). 5 patients did not complete a baseline QOL.
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label-Single Arm
Number analyzed (Participants) | 16
Participants
  Showed overall improvement in mean QOL from baseline | 7
  Showed no change in mean QOL from baseline | 4
  Showed overall decrease in mean QOL from baseline | 5

ADVERSE EVENTS:
Time Frame: All adverse events (AE's), and deaths recorded from initiation of investigational product (IP), until 30 days of the last study intervention, should be followed to their resolution, or until the investigator assesses them as stable, determines the event to be irreversible, or the participant is lost to follow-up. AE's will be recorded for each patient, from the first day of treatment with IP until 30 days after the last dose of IP. Approximately up to 1840 days.
Arm/Group | Open Label-Single Arm
All-Cause Mortality (participants affected / at risk) | 2/22
Serious Adverse Events (participants affected / at risk) | 17/22
Other Adverse Events (participants affected / at risk) | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label-Single Arm (N=22)
Nausea (Gastrointestinal disorders) | 1 (1) — Grade 3
Right hand MSSA cellulitis (General disorders) | 1 (1) — Grade 3
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) — Grade 3
Cellulitis (General disorders) | 1 (1) — Grade 4
Atrial fibrillation (Cardiac disorders) | 1 (1) — Grade 3
Chronic lymphocytic leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Grade 3
COVID-19 infection (Infections and infestations) | 1 (1) — Grade 5
Delirium (General disorders) | 1 (1) — Grade 3
Dyspnea (General disorders) | 1 (1) — Grade 3
E.Coli Sepsis (Infections and infestations) | 1 (1) — Grade 4
Fall (General disorders) | 1 (1) — Grade 3
Fatigue (General disorders) | 1 (1) — Grade 2
Fever (General disorders) | 2 (2) — Grade 3
Gastrointestinal bleed (Blood and lymphatic system disorders) | 1 (1) — Grade 3
Legionella pnemonia (Infections and infestations) | 1 (1) — Grade 3
Myositis (Skin and subcutaneous tissue disorders) | 1 (1) — Grade 3
Peripheral ischemia (Blood and lymphatic system disorders) | 1 (1) — Grade 3
Platelet transfusion reaction (General disorders) | 1 (1) — Grade 3
Pneumonia (Infections and infestations) | 1 (1) — Grade 5
Progression to AML (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Grade 5
Salmonella diarrhea (Infections and infestations) | 1 (1) — Grade 3
Severe anemia (Blood and lymphatic system disorders) | 1 (1) — Grade 3
Splenic pain (General disorders) | 1 (1) — Grade 3
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) — Grade 4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label-Single Arm (N=22)
Abdominal cramping (Gastrointestinal disorders) | 2 (2) — Grade 1
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) — Grade 2
Abdominal pain (Gastrointestinal disorders) | 4 (6) — Grade 1/2
Anorexia (General disorders) | 3 (3) — Grade 2
Appetite change (General disorders) | 6 (13) — Grade 1
Back pain (General disorders) | 4 (4) — Grade 1
Edema (Blood and lymphatic system disorders) | 5 (16) — Grade 1/2
Bone/joint pain (Musculoskeletal and connective tissue disorders) | 13 (14) — Grade 1/2
Bruising/bleeds easily (Blood and lymphatic system disorders) | 5 (11) — Grade 1
Calf cramps/pain (Musculoskeletal and connective tissue disorders) | 3 (3) — Grade 1
Mouth sores (Skin and subcutaneous tissue disorders) | 4 (7) — Grade 1/Grade 2
Chills/rigors (General disorders) | 6 (8) — Grade 1/2
Congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Grade 2
Constipation (Gastrointestinal disorders) | 9 (11) — Grade 1/2
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (11) — Grade 1/2
Diaphoresis (General disorders) | 2 (2) — Grade 1
Diarrhea (Gastrointestinal disorders) | 8 (13) — Grade 1/2
Diffuse achiness (General disorders) | 2 (3) — Grade 1
Dizziness (Nervous system disorders) | 9 (23) — Grade 1/2
Dry mouth (General disorders) | 2 (2) — Grade 1
Dyspnea (Reproductive system and breast disorders) | 10 (19) — Grade 1/2/3
Dysuria (Renal and urinary disorders) | 2 (2) — Grade 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 (8) — Grade 1
Fall (General disorders) | 2 (4) — Grade 1/2
Fatigue (General disorders) | 15 (34) — Grade 1/2/3
Fecal urgency (Gastrointestinal disorders) | 2 (2) — Grade 1
Fever (General disorders) | 4 (5) — Grade 1/2
Headache (General disorders) | 6 (7) — Grade 1/2
Hemangioma (Blood and lymphatic system disorders) | 2 (2) — Grade 1
Hemorrhagic bullae (Skin and subcutaneous tissue disorders) | 2 (5) — Grade 1/2
Hypocalcemia (Metabolism and nutrition disorders) | 2 (6) — Grade 2
Itching (Skin and subcutaneous tissue disorders) | 4 (4) — Grade 1/2
Muscle cramps (Musculoskeletal and connective tissue disorders) | 2 (2) — Grade 1/2
Nausea (Gastrointestinal disorders) | 8 (19) — Grade 1/2
Night sweats (General disorders) | 5 (5) — Grade 1/2
Pneumonia (Infections and infestations) | 2 (2) — Grade 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) — Grade 1/2
Pallor (General disorders) | 5 (8) — Grade 1
Splenomegaly (General disorders) | 3 (3) — Grade 1
Palpitations (Cardiac disorders) | 2 (3) — Grade 1/2
Petechiae (Skin and subcutaneous tissue disorders) | 4 (4) — Grade 1
Progression to AML (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 4 (4) — Grade 1
Shoulder pain (General disorders) | 3 (5) — Grade 1/2
Sore throat (General disorders) | 3 (3) — Grade 1
Upper respiratory infection (Infections and infestations) | 2 (2) — Grade 1
Weakness (General disorders) | 6 (6) — Grade 1/2
Weight loss (General disorders) | 3 (3) — Grade 2
Wheezes (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Grade 1
Anemia (Blood and lymphatic system disorders) | 17 (47) — Grade 3

LIMITATIONS AND CAVEATS:
The statistical analysis plan (and associated statistical power) was based on an expected sample size of 47 evaluable patients. Forty-six patients were consented and ultimately only 16 patients were evaluable. This reduced sample size was not sufficient for the statistical analysis plan as written, and, therefore, only descriptive statistics for the response proportions can be presented for the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-22): https://cdn.clinicaltrials.gov/large-docs/26/NCT03075826/Prot_SAP_000.pdf